CLINICAL TRIAL: NCT04551196
Title: Effectiveness of a Combined Acetaminophen and Ibuprofen Regimen for Management of Post-Tonsillectomy Pain in Pediatric Patients
Brief Title: Management of Post-Tonsillectomy Pain in Pediatric Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202002118
Record Dates: First submitted 2020-09-09; First posted 2020-09-16 (Actual); Results first posted 2024-07-11 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Pain, Postoperative; Tonsillar Hypertrophy; Tonsillitis
MeSH Terms: conditions — Pain, Postoperative; Tonsillitis | interventions — Ibuprofen

STUDY DESIGN:
Intervention Model Description: Single-center, randomized, open-label, non-inferiority treatment pilot study
Masking Description: Open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Alternating Regimen (Active Comparator): A regimen of acetaminophen and ibuprofen alternating doses every 3 hours.
  Interventions: Drug: Alternating Acetaminophen and Ibuprofen
- Combined Regimen (Active Comparator): A regimen of acetaminophen and ibuprofen dosed together every 6 hours.
  Interventions: Drug: Combined Acetaminophen and Ibuprofen

INTERVENTIONS:
Drug: Alternating Acetaminophen and Ibuprofen — Subjects will alternate their post-operative acetaminophen and ibuprofen every 3 hours.
  Other Names: Alternating regimen
  Arms: Alternating Regimen
Drug: Combined Acetaminophen and Ibuprofen — Subjects will take their post-operative acetaminophen and ibuprofen together every 6 hours.
  Other Names: Combined regimen
  Arms: Combined Regimen

SUMMARY:
Single-center, randomized, open-label, non-inferiority treatment pilot study to evaluate the effectiveness of a combined acetaminophen and ibuprofen regimen for treatment of post-operative tonsillectomy pain in the pediatric population. 100 children undergoing tonsillectomy will be randomized to receive either a combined acetaminophen and ibuprofen regimen dosed every 6 hours or an alternating regimen of acetaminophen and ibuprofen dosed every 3 hours.

ELIGIBILITY:
Inclusion Criteria:

* 4 to 17 years of age at time of enrollment
* Undergoing tonsillectomy with or without adenoidectomy
* Able to provide informed consent from parent or legal guardian
* Able to provide assent if subject is a minor of appropriate age

Exclusion Criteria:

* Allergy to acetaminophen or ibuprofen
* Inability for study participant to cooperate with pain assessments
* Known pregnancy
* Any condition which would make the participant, in the opinion of the investigator, unsuitable for the study

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2020-09-28 (Actual); Primary Completion 2022-11-10 (Actual); Study Completion 2022-11-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Louis Children's Hospital, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mitchell RB, Archer SM, Ishman SL, Rosenfeld RM, Coles S, Finestone SA, Friedman NR, Giordano T, Hildrew DM, Kim TW, Lloyd RM, Parikh SR, Shulman ST, Walner DL, Walsh SA, Nnacheta LC. Clinical Practice Guideline: Tonsillectomy in Children (Update). Otolaryngol Head Neck Surg. 2019 Feb;160(1_suppl):S1-S42. doi: 10.1177/0194599818801757. PMID 30798778
- [Background] Ingram DG, Friedman NR. Toward Adenotonsillectomy in Children: A Review for the General Pediatrician. JAMA Pediatr. 2015 Dec;169(12):1155-61. doi: 10.1001/jamapediatrics.2015.2016. PMID 26436644
- [Background] National Prospective Tonsillectomy Audit Final Report. Royal College of Surgeons https://www.rcseng.ac.uk/library-and-publications/rcs-publications/docs/tonsillectomy-audit/
- [Background] Alvarez Palacios I, Gonzalez-Orus Alvarez-Morujo R, Alonso Martinez C, Ayala Mejias A, Arenas Britez O. Postoperative Pain in Adult Tonsillectomy: Is There Any Difference Between the Technique? Indian J Otolaryngol Head Neck Surg. 2017 Jun;69(2):187-193. doi: 10.1007/s12070-017-1058-9. Epub 2017 Jan 16. PMID 28607888
- [Background] Lauder G, Emmott A. Confronting the challenges of effective pain management in children following tonsillectomy. Int J Pediatr Otorhinolaryngol. 2014 Nov;78(11):1813-27. doi: 10.1016/j.ijporl.2014.08.011. Epub 2014 Aug 27. PMID 25241379
- [Background] Tobias JD, Green TP, Cote CJ; SECTION ON ANESTHESIOLOGY AND PAIN MEDICINE; COMMITTEE ON DRUGS. Codeine: Time to Say "No". Pediatrics. 2016 Oct;138(4):e20162396. doi: 10.1542/peds.2016-2396. Epub 2016 Sep 19. PMID 27647717
- [Background] Kelly LE, Sommer DD, Ramakrishna J, Hoffbauer S, Arbab-Tafti S, Reid D, Maclean J, Koren G. Morphine or Ibuprofen for post-tonsillectomy analgesia: a randomized trial. Pediatrics. 2015 Feb;135(2):307-13. doi: 10.1542/peds.2014-1906. PMID 25624387
- [Background] Ismail Zaidan & Amanda Lent. Post-Tonsillectomy Pain in Children: The Postcodeine Era. US Pharm. 41, 31-34 (2016).
- [Background] D'Souza JN, Schmidt RJ, Xie L, Adelman JP, Nardone HC. Postoperative nonsteroidal anti-inflammatory drugs and risk of bleeding in pediatric intracapsular tonsillectomy. Int J Pediatr Otorhinolaryngol. 2015 Sep;79(9):1472-6. doi: 10.1016/j.ijporl.2015.05.042. Epub 2015 Jul 2. PMID 26164211
- [Background] Lewis SR, Nicholson A, Cardwell ME, Siviter G, Smith AF. Nonsteroidal anti-inflammatory drugs and perioperative bleeding in paediatric tonsillectomy. Cochrane Database Syst Rev. 2013 Jul 18;2013(7):CD003591. doi: 10.1002/14651858.CD003591.pub3. PMID 23881651
- [Background] Merry AF, Gibbs RD, Edwards J, Ting GS, Frampton C, Davies E, Anderson BJ. Combined acetaminophen and ibuprofen for pain relief after oral surgery in adults: a randomized controlled trial. Br J Anaesth. 2010 Jan;104(1):80-8. doi: 10.1093/bja/aep338. PMID 20007794
- [Background] Miranda HF, Puig MM, Prieto JC, Pinardi G. Synergism between paracetamol and nonsteroidal anti-inflammatory drugs in experimental acute pain. Pain. 2006 Mar;121(1-2):22-8. doi: 10.1016/j.pain.2005.11.012. Epub 2006 Feb 9. PMID 16480830
- [Background] Gardiner P, Dvorkin L. Promoting medication adherence in children. Am Fam Physician. 2006 Sep 1;74(5):793-8. PMID 16970023
- [Background] Haynes RB, McKibbon KA, Kanani R. Systematic review of randomised trials of interventions to assist patients to follow prescriptions for medications. Lancet. 1996 Aug 10;348(9024):383-6. doi: 10.1016/s0140-6736(96)01073-2. PMID 8709739
- [Background] Uitti JM, Salantera S, Laine MK, Tahtinen PA, Ruohola A. Adaptation of pain scales for parent observation: are pain scales and symptoms useful in detecting pain of young children with the suspicion of acute otitis media? BMC Pediatr. 2018 Dec 20;18(1):392. doi: 10.1186/s12887-018-1361-y. PMID 30572868

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible candidates scheduled to undergo tonsillectomy at SLCH were approached either in the outpatient setting or preoperative holding area prior to surgery by the study team. Recruitment period was from 3/2020 - 10/2021.
Period: Overall Study
Arm/Group | Alternating Regimen | Combined Regimen
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Alternating Regimen | Combined Regimen | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 25 | 25 | 50
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 10 | 26
  Male | 9 | 15 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 25 | 23 | 48
  Unknown or Not Reported | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 4 | 8
  White | 21 | 20 | 41
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With FLACC Pain Scores ≥7 From POD 1 Through POD 3
Description: The proportion of FLACC (Faces, Legs, Activity, Cry, and Consolability scale) pain scores ≥7 from POD 1 through POD 3 compared between the combined and the alternating medication regimens.
  The FLACC scale is scored in a range of 0-10 with 0 representing no pain. The scale has five criteria (Faces, Legs, Activity, Cry, and Consolability), which are each assigned a score of 0, 1 or 2.
Time Frame: up to 3 days following consent
Measure: Number; unit: participants
Arm/Group | Alternating Regimen | Combined Regimen
Number analyzed (Participants) | 25 | 25
participants | 1 | 1

2. Secondary Outcome: Number of Participants With FLACC Pain Scores ≥7 on Each Individual POD 1, 3, and 7
Description: The proportion of FLACC (Faces, Legs, Activity, Cry, and Consolability scale) pain scores ≥7 on each individual POD 1, 3, and 7 compared between the combined and the alternating medication regimens.
  The FLACC scale is scored in a range of 0-10 with 0 representing no pain. The scale has five criteria (Faces, Legs, Activity, Cry, and Consolability), which are each assigned a score of 0, 1 or 2.
Time Frame: 3 separate individual days, will be completed days after the surgery
Measure: Number; unit: participants
Arm/Group | Alternating Regimen | Combined Regimen
Number analyzed (Participants) | 25 | 25
participants | 1 | 1

3. Secondary Outcome: Number of Participants With FLACC Pain Scores ≥7 From POD 1 Through POD 7
Description: The proportion of cumulative FLACC pain scores ≥7 from POD 1 through POD 7 compared between the combined and the alternating medication regimens.
  The FLACC scale is scored in a range of 0-10 with 0 representing no pain. The scale has five criteria (Faces, Legs, Activity, Cry, and Consolability), which are each assigned a score of 0, 1 or 2.
Time Frame: up to 7 days following consent
Measure: Number; unit: participants
Arm/Group | Alternating Regimen | Combined Regimen
Number analyzed (Participants) | 25 | 25
participants | 1 | 1

4. Secondary Outcome: Number of Participants With Faces Pain Scores ≥8 on POD 1, 3, and 7
Description: The proportion of Faces pain scores ≥8 on POD 1, 3, and 7 compared between the combined and the alternating medication regimens.
  The Faces scale shows a series of faces ranging from a happy face at 0, or "no hurt", to a crying face at 10, which represents "hurts like the worst pain imaginable". Based on the faces and written descriptions, the patient chooses the face that best describes their level of pain.
Time Frame: 3 separate individual days, will be completed days after the surgery
Measure: Number; unit: participants
Arm/Group | Alternating Regimen | Combined Regimen
Number analyzed (Participants) | 25 | 25
participants | 1 | 1

5. Secondary Outcome: Number of Participants With Cumulative Faces Pain Scores ≥8 From POD 1 Through POD 7
Description: The proportion of cumulative Faces pain scores ≥8 from POD 1 through POD 7 compared between the combined and the alternating medication regimens.
  The Faces scale shows a series of faces ranging from a happy face at 0, or "no hurt", to a crying face at 10, which represents "hurts like the worst pain imaginable". Based on the faces and written descriptions, the patient chooses the face that best describes their level of pain.
Time Frame: up to 7 days following consent
Measure: Number; unit: participants
Arm/Group | Alternating Regimen | Combined Regimen
Number analyzed (Participants) | 25 | 25
participants | 3 | 1

6. Secondary Outcome: Number of Participants With Rescue Medication Usage Through POD 3
Description: The proportion of rescue medication usage from POD 1 through POD 3 compared between the combined and the alternating medication regimens.
Time Frame: up to 3 days following consent
Measure: Number; unit: participants
Arm/Group | Alternating Regimen | Combined Regimen
Number analyzed (Participants) | 25 | 25
participants | 3 | 7

7. Secondary Outcome: Number of Participants With Rescue Medication Usage Through POD 7
Description: The proportion of rescue medication usage from POD 1 through POD 7 compared between the combined and the alternating medication regimens.
Time Frame: up to 7 days following consent
Measure: Number; unit: participants
Arm/Group | Alternating Regimen | Combined Regimen
Number analyzed (Participants) | 25 | 25
participants | 1 | 0

8. Secondary Outcome: Proportion of Subjects That Adhere to the Assigned Medication Regimen
Description: Proportion of subjects that adhere to the assigned medication regimen compared between the combined and the alternating medication regimens as determined by the medication log that the participants return at the end of the study.
Time Frame: up to 3 days following consent
Measure: Count of Participants; unit: Participants
Arm/Group | Alternating Regimen | Combined Regimen
Number analyzed (Participants) | 25 | 25
Participants | 25 | 25

9. Secondary Outcome: Adverse Events
Description: Incidence of adverse events
Time Frame: up to 7 days following consent
Population: Alternating regimen
Measure: Number; unit: participants
Arm/Group | Alternating Regimen | Combined Regimen
Number analyzed (Participants) | 25 | 25
participants | 3 | 3

ADVERSE EVENTS:
Time Frame: Adverse event data was collected post operatively days 1 through 7
Description: Follow up surveys to assess pain scores and adverse events were sent to participants twice a day on post-operative day (POD) 1, 3, and 7.
Arm/Group | Alternating Regimen | Combined Regimen
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 3/25 | 3/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alternating Regimen (N=25) | Combined Regimen (N=25)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Emesis (Gastrointestinal disorders) | 3 (3) | 1 (1)
Bloody Oral Secretions (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pain - Uncontrolled (General disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-02-10): https://cdn.clinicaltrials.gov/large-docs/96/NCT04551196/Prot_SAP_ICF_005.pdf